CLINICAL TRIAL: NCT04537273
Title: Clinical and Pathological Characteristics as Prognostic Factors in Locally Advanced Cervical Cancer: A Retrospective Study
Brief Title: Clinical and Pathological Characteristics as Prognostic Factors in Locally Advanced Cervical Cancer
Status: Completed | Type: Observational
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Principal Investigator, David Cantu, Md, PhD, National Institute of Cancerología
Other Study IDs: Rev/050/18
Record Dates: First submitted 2020-08-25; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Cervical Cancer
Keywords: Locally advanced; Cervical carcinoma; Prognostic factors
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Localy advanced Cervical Cancer: Patients with Localy advanced Cervical Cancer confirmed by pathology, clinical exams and computed tomography scan, treated with concurrent chemoradiotherapy.
  Interventions: Other: Descriptive and analytical

INTERVENTIONS:
Other: Descriptive and analytical

SUMMARY:
Locally advanced cervical cáncer continues to be a public health problem in emergent economies, even though treatment is very well standardized, recurrence rate is still high, making necessary to evaluate prognostic clinical and pathological factors. The aim of this study is to evaluate clinical and pathological prognostic factor in terms of treatment outcomes, disease-free survival (DFS) and overall survival (OS) in a retrospective cohort of patients with LACC treated with standard chemoradiotherapy in a reference center in México.

DETAILED DESCRIPTION:
This is a retrospective study, the data were obtained from clinical files of cervical cancer patients with clinical stages IB2-IVA(FIGO2009) treated at the Instituto Nacional de Cancerología in Mexico City from January 2005 to December 2014.

A total of 1954 patients with LACC confirmed by pathology, clinical exams and computed tomography scan (CT) were identified.

Demographic, clinical, pathological and follow-up as well as survival status of all patients was recorded. Treatment outcome was classified as complete response if the patient had no signs of tumor activity after 6 months of finishing treatment, persistence of disease was defined if tumor could be identified after treatment or before six months of treatment termination, progression was defined if tumor growth occurred or metastatic disease appeared. Disease-free survival (DFS) was defined as the period between finishing treatment and the occurrence of relapse, which was confirmed by pathological study and/or CT. Overall survival (OS) was defined as the time period between diagnosis and death or date at last visit. Quantitative variables were described with central tendency and dispersion measures and analyzed with Student's t or Mann-Whitney U test. Normality was determined with Shapiro-Wilk's test, Chi-squared for categorical comparisons between groups, Kaplan-Meir with the log-rank test for survival analysis were performed. The multivariate analysis was performed using Cox proportional Hazard regression model. Statistically significant differences were defined as a p value <0.05.

Statistical analyses were performed using IBM SPSS, version 23 (IBM Corp., Armonk, N.Y., USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with cervical cancer clinical stage Ib2-IVa
* Treated with concomitant Chemoradiotherapy

Exclusion Criteria:

* Rare histologies such gastric type adenocarcinoma, neuroendocrine or clear-cell carcinoma
* incomplete treatment or not treated with chemoradiotherapy
* Two primary malignancies
* Insufficient data for analysis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Locally advanced cervical cancer confirmed by pathology, clinical exams and computed tomography scan (CT)
Sampling Method: Non-Probability Sample
Enrollment: 1954 (Actual)
Dates: Start 2005-01-02 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Analyze the clinical and pathological characteristics as prognostic factor of patients with locally advanced cervical cancer. | 5 years
  Analyze the clinical and pathological characteristics of patients with cervical cancer stages IB2 to IVA as prognostic factor in terms of overall survival.

SECONDARY OUTCOMES:
Analyze the clinical and pathological characteristics as prognostic factor of patients with locally advanced cervical cancer. | 6 months
  Analyze the clinical and pathological characteristics of patients with cervical cancer stages IB2 to IVA as prognostic factor in terms of response rate of treatment.
Analyze the clinical and pathological characteristics as prognostic factor of patients with locally advanced cervical cancer. | 5 years
  Analyze the clinical and pathological characteristics of patients with cervical cancer stages IB2 to IVA as prognostic factor in terms of disease-free survival.

IPD SHARING:
Plan to Share IPD: Yes
Direct request to the principal investigator
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Any time by direct request to the principal investigator
Access Criteria: Only for research purpose.

REFERENCES:
- [Derived] Gallardo-Alvarado L, Cantu-de Leon D, Ramirez-Morales R, Santiago-Concha G, Barquet-Munoz S, Salcedo-Hernandez R, Reyes C, Perez-Alvarez S, Perez-Montiel D, Perez-Plasencia C, Trejo-Duran E, Galicia JP. Tumor histology is an independent prognostic factor in locally advanced cervical carcinoma: A retrospective study. BMC Cancer. 2022 Apr 13;22(1):401. doi: 10.1186/s12885-022-09506-3. PMID 35418030